CLINICAL TRIAL: NCT05551923
Title: Predictive Value of Human Microbiome and Serological Markers for Clinical Outcome of Cerebral Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-168
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Hemorrhagic Stroke; Acute; Outcomes; Metabolites; Gut Microbiota
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, oral swabs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute cerebral hemorrhage: intestinal flora disturbance To observe the clinical prognosis of acute cerebral hemorrhage after enterobacterial disorder
  Interventions: Other: intestinal flora disturbance
- The group without stroke: The group without stroke

INTERVENTIONS:
Other: intestinal flora disturbance — To observe the clinical prognosis of acute cerebral hemorrhage after enterobacterial disorder
  Groups: Acute cerebral hemorrhage

SUMMARY:
Objective: To explore the predictive value of characteristic disorder of intestinal flora for clinical prognosis in patients with intracerebral hemorrhage. Secondary objectives: 1) To investigate the correlation of gut microbiota and its serological indicators with imaging features and clinical neurological deficits in ICH; 2) Dynamically observe the changes of human microbiome and its serological indicators after ICH, and explore the biomarkers based on human microbiome related to disease changes.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage has brought a heavy burden to society and families. Finding biomarkers closely related to the condition of intracerebral hemorrhage is an important research direction for the prevention and treatment of intracerebral hemorrhage. However, there are few studies on the correlation between cerebral hemorrhage and microbiota. Our previous small sample study found that there were intestinal flora and SCFAs metabolism disorders in patients with hypertensive cerebral hemorrhage, and the latter was significantly related to poor prognosis. These results suggest that gut microbiota and its metabolites may become prognostic predictors and therapeutic targets for patients with intracerebral hemorrhage. However, more research evidence is still needed to confirm. Therefore, this study hypothesized that oral or intestinal flora in patients with acute cerebral hemorrhage has a certain degree of disorder and dynamic changes, accompanied by changes in serum markers, and there is a potential relationship between the changes of some microbiota-related markers and the severity and outcome of cerebral hemorrhage. Therefore, this topic proposed collection in patients with acute cerebral hemorrhage oral swabs, blood and feces or anal swab specimens, evaluate the neurological function score, imaging features and clinical outcomes, and to establish a follow-up queue, the dynamic change of cerebral hemorrhage patients after intestinal bacterial flora and condition and poor prognosis, the correlation of biomarkers new prediction and prevention of brain hemorrhage, To improve the effectiveness of prevention and treatment of cerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. It meets the diagnostic criteria for acute ischemic stroke
2. Age ≥ 18 years
3. The onset time is less than or equal to 2 weeks
4. Diagnosis of cancer before stroke onset or during hospitalization and active cancer (failure to meet clinical criteria for cure, or discovery of recurrence or metastasis)
5. Sign an informed consent form, provide relevant medical history information and provide biological specimens

Exclusion Criteria:

1. Previous history of disabling stroke (pre-onset mRS ≥2)
2. Primary central nervous system tumor or hematologic system tumor
3. The cancer meets the criteria for clinical cure and has not recurred or metastasized for more than 5 years
4. Antibiotics, prebiotics/probiotics taken within 1 month
5. Patients who cannot have stool specimens within 4 days of admission

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute hemorrhagic stroke
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Neurological function score (mRS score) | 3 months after onset
  Neurological function score (mRS score)
mortality | within 12 months after onset
  mortality

SECONDARY OUTCOMES:
New cerebrovascular events | within 12 months after onset
  Occurrence of ischemic stroke and hemorrhagic stroke
NIHSS | The first day and the seventh day after admission, 3 months, 6 months and 12 months after onset
  NIHSS
Barthel Index | 3 months, 6 months and 12 months after onset
  BI
Mini-mental State Examination | The first day and the seventh day after admission, 3 months and 6 months after onset
  MMSE
Montreal Cognitive Assessment | The first day and the seventh day after admission、3 months and 6 months after onset
  MOCA

CONTACTS AND LOCATIONS:
Overall Officials: JIA YIN, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- JIA YIN, Guangzhou, Guangdong, China